CLINICAL TRIAL: NCT01504906
Title: A Single-Center,Open-Label,Randomized,3-Treatment,3-Period Cross-Over Study to Investigate the Potential Effect of Cyclosporine on the Pharmacokinetics, Safety, and Tolerability of Ticagrelor and the Effect of Ticagrelor on the Pharmacokinetics, Safety, and Tolerability of Cyclosporine
Brief Title: Study to Assess Effect of Cyclosporine on the Blood Levels of Ticagrelor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5130C00074
Record Dates: First submitted 2012-01-02; First posted 2012-01-06 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Phase 1; Healthy male volunteers; pharmacokinetics; cyclosporine; ticagrelor; Bioavailability (plasma AUC, Cmax, plasma AUC0-t, t1/2λz, tmax)
MeSH Terms: interventions — Cyclosporine; Ticagrelor

ARMS (3):
- A (Experimental): cyclosporine 600 mg+ a single oral dose of 180 mg ticagrelor
  Interventions: Drug: cyclosporine; Drug: ticagrelor
- B (Experimental): single dose cyclosporine 600 mg
  Interventions: Drug: cyclosporine
- C (Experimental): single dose 180 mg ticagrelor
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: cyclosporine — Oral tablets, 600 mg , single dose
  Arms: A; B
Drug: ticagrelor — Oral tablets, 180 mg, single dose
  Arms: A; C

SUMMARY:
The purpose of this study is to assess the effect of Cyclosporine on the blood levels of Ticagrelor.

DETAILED DESCRIPTION:
A Single-Center,Open-Label,Randomized,3-Treatment,3-Period Cross-Over Study to Investigate the Potential Effect of Cyclosporine on the Pharmacokinetics, Safety, and Tolerability of Ticagrelor and the Effect of Ticagrelor on the Pharmacokinetics, Safety, and Tolerability of Cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent prior to any study-specific procedures
* Healthy male subjects aged 18 to 45 years (inclusive) with suitable veins for cannulation or repeated venipuncture

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* A history of hemophilia, von Willebrand's disease, lupus anti-coagulant, or other diseases/syndromes that can either alter or increase the propensity for bleeding
* A personal history of vascular abnormalities including aneurysms; a personal history of severe hemorrhage, hematemesis, melena, hemoptysis, severe epistaxis, severe thrombocytopenia, intracranial hemorrhage, or rectal bleeding within 1 year

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetic (PK) profile for Ticagrelor and its metabolite AR-C124910XX in terms of maximum concentration (Cmax),time to maximum concentration (tmax) and area under the concentration curve from time zero to infinity (AUC) | PK samples will be collected postdose 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, and 48 hours
  PK samples will be collected postdose at visits 2,3 and 4
Description of the PK profile for Ticagrelor and its metabolite AR-C124910XX in terms of area under the concentration-time curve from time zero to the last measurable concentration (AUC(0-t)),terminal half-life (t1/2) | PK samples will be collected postdose 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, and 48 hours
  PK samples will be collected postdose at visit 2,3 and 4
Description of the PK profile for AR-C124910XX : ticagrelor in terms of ratios for Cmax, AUC(0-t), and AUC | PK samples will be collected postdose 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, and 48 hours
  PK samples will be collected postdose at visit 2,3 and 4
Description of the PK profile for Cyclosporine in terms of Cmax, AUC(0-t), AUC, tmax and t1/2 | PK samples will be collected postdose 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, and 48 hours
  PK samples will be collected postdose at visit 2,3 and 4

SECONDARY OUTCOMES:
Description of the safety profile in terms of adverse events, blood pressure, pulse, temperature, ECG (Electrocardiogram), physical examination, and safety laboratory variables | Baseline up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Miriana Kujacic, MD, Study Chair — Molndal, Sweden AstraZeneca; Kelli Craven, MD, Principal Investigator — Overland Park US, Quintiles, Inc.
Locations (1):
- Research site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Teng R, Kujacic M, Hsia J. Pharmacokinetic interaction study of ticagrelor and cyclosporine in healthy volunteers. Clin Drug Investig. 2014 Aug;34(8):529-36. doi: 10.1007/s40261-014-0205-2. PMID 24861133